CLINICAL TRIAL: NCT00219973
Title: Multicentric, Rand., D-b, Pbo Controlled Clinical Trial to Evaluate the Efficacy and the Safety of the Thromboprophylaxis With Bemiparin 3,500 IU/d for 28 Days Compared to 8 Days, in Patients Undergoing Oncological Abdominal/ Pelvic Surgery
Brief Title: CANBESURE STUDY (Cancer, Bemiparin and Surgery Evaluation)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ROV-BEM-2003-02
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Cancer; Venous Thromboembolism
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary embolism; bleeding; low-molecular-weight heparin; cancer; surgery
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Hemorrhage | interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bemiparin — Bemiparin 3.500 IU/day for 28 days compared to 8 days

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of Bemiparin, a second-generation LMWH, in the prophylaxis of VTE (using a postoperative regimen, i.e. administering the first dose 6 hours after finishing the surgical procedure) for 28 days compared to 8 days, in oncological surgery.

DETAILED DESCRIPTION:
Although the efficacy of low-molecular-weight heparins(LMWH) in the prophylaxis of postoperative venous thromboembolism (VTE) is well established in a large number of studies, some aspects remain to be determined. The optimal duration of prophylactic treatment has not been clearly defined yet.

Traditionally, surgical prophylaxis of VTE in patients undergoing high-risk orthopaedic surgery was extended for one or two weeks after the operation. However, the most recent studies carried out on this field have demonstrated that prolongation of prophylaxis with LMWH for 4-6 weeks significantly reduces the incidence of VTE (by more than half) in patients undergoing orthopaedic surgery with a high-risk of VTE.

On the contrary, thromboprophylaxis in oncological surgery is generally limited to the period of hospitalisation, despite the fact that activation of coagulation is greater and more prolonged in patients undergoing surgery for neoplastic processes than in those patients not affected by cancer. The only two studies carried out to evaluate the efficacy of the prolongation of thromboprophylaxis for 4 weeks in this type of surgery seem to indicate that the VTE incidence could be reduced even further that with one-week prophylaxis, though these do not allow to establish a definitive conclusion.

The present study aims to evaluate the efficacy and safety of Bemiparin, a second-generation LMWH, in the prophylaxis of VTE (using a postoperative regimen, giving the first dose 6 hours after finishing the surgical procedure) for 28 days compared to 8 days, in oncological surgery.

Additionally, some exploratory analyses will be carried out to evaluate:

1. The biological effect of the sc. administration of Bemiparin (3,500 IU/day) on different biological markers involved in the tumoral development and its metastasis in patients undergoing an oncological abdominal or pelvic surgical operation.
2. The effect of the sc. administration of Bemiparin (3,500 IU/day) on the evolution of the tumour in patients undergoing an oncological abdominal or pelvic surgical operation.
3. The effect of the sc. administration of Bemiparin (3,500 IU/day) on the survival of the patients at 6 months from the operation.

Four Study Committees have been created for this clinical trial in order to guarantee the safety of the patients as well as the highest quality data:

* Trial Steering Committee
* Data & Safety Monitoring Board
* Committee for the Evaluation of Phlebographies
* Committee for Adjudicating Clinical Events.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 40 years of age or older, of either sex, who have given their informed consent to participate in the study.
* Patients with a malignant neoplastic process (primary or metastasic) of the gastrointestinal tract (except the oesophagus), genitourinary tract or female reproductive organs, previously diagnosed and documented, and who are programmed to undergo elective, open, curative or palliative surgery directly related to that disease.
* Patients undergoing surgery with general or spinal anaesthesia, with an estimated duration of surgery of over 30 minutes.
* Patients with a life expectancy of at least 3 months.

Exclusion Criteria:

* Curative or palliative surgery of a malignant neoplastic process in liver, biliary tract or pancreas.
* Women who are pregnant or breast-feeding, or women with child-bearing potential who are not using effective contraceptive methods.
* Patients with macrohaematuria, active haemorrhage within the past two months, organ lesions at risk of bleeding (e.g. active peptic ulcer, haemorrhagic cerebrovascular accident, aneurysms), a history of episodes of clinically evident haemorrhage, major surgery in the previous month or an increase in the risk of bleeding due to any disturbance of haemostasis which would contraindicate the anticoagulant therapy, with the exception of bleedings episodes directly caused by tumour subjected to the surgical intervention.
* Patients with known hypersensitivity to the LMWHs, to heparin or to substances of porcine origin.
* Patients with known hypersensitivity to radiological contrast media.
* Patients with known hypersensitivity to anaesthetic drugs or pre-anaesthetic drugs.
* Patients with a congenital or acquired bleeding diathesis (confirmed by hematological test), with or without haematuria.
* Lesions or surgical interventions of the central nervous system, eyes or ears within the previous 6 months, including hemorrhagic or ischemic cerebro-vascular accident, cerebral thrombosis and/or known cerebral metastasis.
* Disseminated Intravascular Coagulation (DIC) attributable to heparin-induced thrombocytopenia.
* Acute bacterial endocarditis and slow endocarditis.
* Patients on treatment with oral or parenteral anticoagulants within 5 days before the operation.
* Patients with a history of thrombocytopenia associated with heparin or with a current platelet count <75,000/mm3.
* Patients with renal failure (defined as a serum creatinine over 2 mg/dL), hepatic insufficiency (with AST and/or ALT values > 5 times over normal values established by the reference range of the local laboratory of the hospital).
* Severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure over 120 mmHg).
* One or more documented episodes of DVT and/or PE (confirmed by a ventilation-perfusion gamma scan or helical CT) in the previous 3 months.
* Patients with suspected or confirmed inability to comply with the study treatment and/or follow-up.
* Patients who are participating in another clinical trial or who have done so in the past 30 days.
* Patients with a cava vein filter in place.
* Patients needing the use of unallowed concomitant treatments or medications such as more than 125mg/day aspirin, NSAIDs with long half-life of significant anti-aggregation activity, metformin, or any anticoagulant compound (please refer to section of the protocol "Concomitant medications and treatments" for details)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2005-05; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
EFFICACY: Combined incidence (from day 1 to day 20±2 after the randomisation): total DVT + non-fatal PE + all-cause mortality.
SAFETY: incidence of major bleeding (from day 1 to day 20±2 after the randomisation).

SECONDARY OUTCOMES:
EFFICACY: combined and isolated incidence of DVT (Total, proximal and distal), non-fatal PE, deaths related and not related with VTE.
SAFETY: incidence of major bleeding (from day 1 to day 82±8 after the randomisation) and incidence of minor bleeding (from day 1 to day 20±2 and to day 82±8 after the randomisation).
EXPLORATORY ANALYSES: Biological markers, tumour evolution and survival at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay V Kakkar, Prof., Study Director — Thrombosis Research Institute (London, UK); Paolo Prandoni, Prof., Study Director — Faculty of Medicine, University of Padova (Padova, Italy); Jose Luis Balibrea-Cantero, Prof., Study Director — Faculty of Medicine, Complutense University (Madrid, Spain)
Locations (4):
- Lisbon, Portugal
- Timișoara, Romania
- Saint Petersburg, Russia
- Madrid, Spain